CLINICAL TRIAL: NCT05228015
Title: A Phase 1, First-in-Human Study of IK-930, an Oral TEAD Inhibitor Targeting the Hippo Pathway in Subjects with Advanced Solid Tumors
Brief Title: Oral TEAD Inhibitor Targeting the Hippo Pathway in Subjects with Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor strategic reasons
Sponsor: Ikena Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IK930-001
Record Dates: First submitted 2022-01-07; First posted 2022-02-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors, Adult; Solid Tumor; Malignant Pleural Mesothelioma (MPM); Epithelioid Hemangioendothelioma (EHE); NF2 Deficient Mesothelioma; Other NF2 Deficient Solid Tumors and Solid Tumors with YAP1/TAZ Fusion Genes; NF2 Deficiency; YAP1 or TAZ Gene Fusions
Keywords: IK-930; HIPPO Pathway; TEAD; YAP/TAZ; NF2 mutated tumors
MeSH Terms: conditions — Mesothelioma, Malignant; Hemangioendothelioma, Epithelioid | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Part 1 dose escalation: BOIN design; Part 2 dose expansion: 4 parallel cohorts, Simon 2-stage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- IK-930 Single Agent Dose Escalation (Experimental)
  Interventions: Drug: IK-930
- IK-930 Single Agent Dose Expansion (Experimental)
  Interventions: Drug: IK-930
- IK-930 and Osimertinib Combination Dose Escalation (Experimental)
  Interventions: Drug: IK-930; Drug: Osimertinib

INTERVENTIONS:
Drug: IK-930 — tablets for oral administration
Drug: Osimertinib — tablets for oral administration
  Arms: IK-930 and Osimertinib Combination Dose Escalation

SUMMARY:
This is a Phase 1, first-in-human (FIH) clinical study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antitumor activity of IK-930, an oral TEAD inhibitor, administered orally (PO) as monotherapy in subjects with advanced solid tumors with or without gene alterations in the Hippo pathway for whom there are no further treatment options known to confer clinical benefit. The study consists of two phases, an initial Dose Escalation phase followed by a Dose Expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Male or female subjects ≥ 18 years of age.
3. If feasible, subjects must be willing to consent to the submission of formalin-fixed paraffin-embedded tissue blocks or slides of tumor tissue, preferably from pre-treatment, baseline fresh tumor biopsy at Screening. Alternatively, archival tumor FFPE blocks or, unstained slides of tumor tissue from available archival sources are acceptable.
4. In the dose escalation cohort: Subjects with histologically proven advanced, unresectable, locally recurrent, or metastatic malignancy that has progressed on or following standard-of-care therapies and for whom there is no available therapy known to confer clinical benefit, regardless of the presence or absence of NF2 deficiency or other genetic alterations of the Hippo pathway. Subjects with histological confirmation of MPM; subjects with NF2-deficient MPM determined by local test results for testing can also be enrolled as well as subjects with any other solid tumors with documented NF2 deficiency determined by local test results for testing, including, but not limited to, meningioma, cholangiocarcinoma, thymoma, mucoepidermoid NSCLC, HCC, and others. Subjects diagnosed with EHE with documented TAZ-CAMTA1 or YAP1-TFE3 gene fusions, as determined by local tests and subjects with solid tumors who have YAP1/TAZ gene fusions as determined by local test results can also be enrolled in the dose escalation part of the study.
5. In the Dose expansion: Four groups of subjects will be enrolled:

   1. Cohort 1: Subjects with histological confirmed MPM and that have documented NF2 deficiency,
   2. Cohort 2: Subjects with other documented NF2-deficient solid tumors agnostic to tumor type including, but not limited to, meningioma, cholangiocarcinoma, thymoma, NSCLC, HCC, and others.
   3. Cohort 3: Subjects with histopathological diagnosis of epithelioid hemangioendothelioma (EHE) and documented TAZ-CAMTA1 or YAP1-TFE3 gene fusions, as determined by local test results. Subjects who have objective disease progression to prior therapy or have active disease and cancer-related pain requiring narcotics for management are eligible.
   4. Cohort 4: Subjects with any solid tumor with documented YAP1/TAZ gene fusions as determined by local test results.
6. In the Osimertinib Combination Cohort subjects must have a histologically proven, incurable, locally advanced or metastatic NSCLC expressing osimertinib-sensitive EGFR mutations; have evidence of radiological disease progression on prior receipt of Osimertinib and have progressed on additional anticancer therapy such as chemotherapy.
7. Subjects can have measurable or evaluable disease by RECIST 1.1 criteria as assessed by the Investigator/local radiologist.

Exclusion Criteria:

1. Subjects with untreated or symptomatic primary central nervous system (CNS) tumors or with intracranial metastases (excluding primary CNS tumors that may be eligible for enrollment as part of Cohort 2 e.g., NF-2 deficient meningioma)

   a. Subjects with leptomeningeal metastases are excluded
2. Uncontrolled or life-threatening symptomatic concomitant disease
3. Clinically significant cardiovascular disease as defined in the protocol
4. Women who are pregnant or breastfeeding
5. Subjects who are unable to swallow or retain oral medication
6. Prior treatment/exposure to YAP/TAZ/TEAD inhibitors
7. Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of IK-930 | Through study completion, an average of 36 months
  The frequency and severity, incidence of treatment-emergent and treatment-related adverse events using NCI-CTCAE v5.0
Occurrence of Dose Limiting Toxicity during first treatment cycle | Approximately 1 year
RP2D and/or MTD of IK-930 | Approximately 1 year
  Define the recommended phase 2 dose (RP2D) and/or MTD of IK-930

SECONDARY OUTCOMES:
Antitumor activity per RECIST 1.1: Disease control rate (DCR) of IK-930 as a single agent | Through study completion, average of 36 months
Antitumor activity per RECIST 1.1: Time to response (TTR) of IK-930 as a single agent | Through study completion, average of 36 months
Antitumor activity per RECIST 1.1: Duration of response (DOR) of IK-930 as a single agent | Through study completion, average of 36 months
Antitumor activity per RECIST 1.1: Objective response rate (ORR) of IK-930 as a single agent | Through study completion, average of 36 months
Antitumor activity: Median progression-free survival (PFS) of IK-930 as a single agent | Through study completion, average of 36 months
Antitumor activity: Median overall survival (OS) of IK-930 as a single agent | Through study completion, average of 36 months
Pharmacokinetics of IK-930: half-life (t1/2) | Approximately 1 year
Pharmacokinetics of IK-930: Area Under the Curve (AUC) | Approximately 1 year
Pharmacokinetics of IK-930: Maximum Plasma Concentration (Cmax) | Approximately 1 year
Pharmacokinetics of IK-930: Minimum Plasma Concentration (Cmin) | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Kim, MD, Study Director — Ikena Oncology; Caroline Germa, MD, Study Chair — Ikena Oncology
Locations (12):
- United States (9):
  - The University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Start Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Sidney Kimmel Cancer Center at Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas
- Peninsula South Eastern Haematology and Oncology Group (PASO Medical), Frankston, Victoria, Australia
- United Kingdom (2):
  - University Hospitals of Leicester NHS Trust, Leicester, England
  - The Royal Marsden Hospital, London, England

IPD SHARING:
Plan to Share IPD: No